## **Document Coversheet**

Study Title: Clinic to Community Navigation to Improve Diabetes Outcomes

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 3/29/2024 |
| NCT Number: | NCT03474731 |
| IRB Number | 43766 |
| Coversheet created: | 7/3/2024 |

0 ι co IRB Approval 3/29/2024 IRB # 43766 IRB6 CLOSED

IMPORTANT NOTE: You will not be able to change your selections for "Which IRB" and "Protocol Process Type" after saving this section. If you select the wrong IRB or Protocol Process Type, you may need to create a new application.

For guidance, see:

- Which IRB?
- Which Protocol Process Type?
- "Getting Started"

Please contact the Office of Research Integrity (ORI) at 859-257-9428, <a href="mailto:IRBsubmission@uky.edu">IRBsubmission@uky.edu</a>, or <a href="mailto:request a consult">request a consult</a> to resolve any questions prior to saving your selections.

| -Which IRB |
|----------------------------------|
| Medical |
| Protocol Process Type |
| € Exemption |
| Expedited (Must be risk level 1) |
| ଜ Full |

The revised Common Rule expanded exemption certification category 4 for certain secondary research with identifiable information or biospecimens. The regulations no longer require the information or biospecimens to be existing. For more information see the <u>Exemption Categories Tool</u>.

### **PROJECT INFORMATION**

0 unresolved comment(s)

Title of Project: (Use the exact title listed in the grant/contract application, if applicable). If your research investigates any aspect of COVID-19, please include "COVID19" at the beginning of your Project Title and Short Title UK/O Clinic to Community Navigation to Improve Diabetes Outcomes

Short Title Description

Please use a few key words to easily identify your study - this text will be displayed in the Dashboard listing for your study.

A1C

Anticipated Ending Date of Research Project: 1/1/2024

Maximum number of human subjects (or records/specimens to be reviewed) 1400

After approval, will the study be open to enrollment of new subjects or new data/specimen collection? Are you requesting that the UK IRB serve as the lead IRB for a multi-site study, OR that the UK IRB defer review to another IRB? [Click here for "IRB Reliance" help]

Yes a No

If "Yes," before completing your IRB application, fill out the Reliance Request Form and submit it to inbreliance@uky.edu.

RISK LEVEL

0 unresolved comment(s)

-Indicate which of the categories listed below accurately describes this protocol

- (Risk Level 1) Not greater than minimal risk
- ⊂ (Risk Level 3) Greater than minimal risk, no prospect of direct benefit to individual subjects, but likely to yield generalizable knowledge about the subject's disorder or condition.
- $\sim$  (Risk Level 4) Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of subjects.
- \*"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves from those ordinarily encountered in daily life or during the performance of routine physical or psychological examination or tests.
- \*\*\*For Expedited and Exempt Applications, the research activities must be Risk Level 1 (no more than minimal risk to human subjects).\*\*\*

Refer to <u>UK's guidance document</u> on assessing the research risk for additional information.

0 unresolved comment(s)

SUBJECT DEMOGRAPHICS

Age level of human subjects: (i.e., 6 mths.; 2yrs., etc..) 18 to older

### Study Population:

Describe the characteristics of the subject population, including age range, gender, ethnic background and health status. Identify the criteria for inclusion and exclusion.

Provide the following information:

- · A description of the subject selection criteria and rationale for selection in terms of the scientific objectives and proposed study design;
- · A compelling rationale for proposed exclusion of any sex/gender or racial/ethnic group;
- Justification for the inclusion of vulnerable groups such as children, prisoners, adults with impaired consent capacity, or others who may be vulnerable to coercion or undue influence.

Please consider these resources:

**NIH Diversity Policy** 

FDA Diversity Guidance

Adults (age 18+); Appalachian residence, no plans to relocate out of the area in the next 18 months, willingness and ability to participate (i.e., no major cognitive impairment) and HbA1c levels at least 6.5%.

Individuals interested and potentially eligible will be asked to complete human subject protection protocol and verify their blood sugar through HbA1c screening. With the high prevalence of undetected T2DM, interested individuals at elevated risk of T2DM (as determined by the American Diabetes Association Risk Test, with a score of = 2) who have not received a T2DM diagnosis, will be offered HbA1c screening and will be considered eligible if they meet the above criteria. More than one member of a household may participate. We will note such arrangements.

We also will need to recruit health clinics who will allow us to partner with them. We would ask them to allow us to work with their receptionists, or other designated staff member, to help schedule appointments for our participants and receive permission to access participants' EMR. Generally, clinics will be paid \$500 for their participation. We will include clinics that serve our specific participants.

### Attachments

Indicate the targeted/planned enrollment of the following members of minority groups and their subpopulations. Possible demographic sources: Census Regional Analyst Edition, Kentucky Race/Ethnic Table, Kentucky Population Data.

(Please note: The IRB will expect this information to be reported at Continuation Review time for Pre-2019 FDA-regulated Expedited review and Full review applications):

| | Participant Demographics | | | |
|---|---|---|---|---|
| | Cisgender Man 🕡 | Cisgender Woman 🕡 | TGNB/TGE 🕟 | Unknown/Not Reported |
| American<br><b>I</b> ndian/A <b>l</b> askan<br>Native: | 10 | 15 | | |
| Asian: | 5 | 10 | | |
| B <b>l</b> ack/African<br>American: | 60 | 70 | | |
| Latinx: | 5 | 10 | | |
| Native<br>Hawaiian/Pacific<br><b>I</b> s <b>l</b> ander: | | | | |
| White: | 515 | 690 | | |
| American<br>Arab/Midd <b>l</b> e<br>Eastern/North<br>African: | | | | |
| Indigenous<br>People Around<br>the World: | | | | |
| More than One<br>Race: | | | | |
| Unknown or Not Reported: | 5 | 5 | | |

### If unknown, please explain why:

Adults (age 18+); Appalachian residence, no plans to relocate out of the area in the next 18 months, willingness and ability to participate (i.e., no major cognitive impairment) and HbA1c levels at least 6.5%.

Indicate the categories of subjects and controls to be included in the study. You may be required to complete additional forms depend the subject categories which apply to your research. If the study does not involve direct intervention or direct interaction with subjects, record-review research, outcomes registries), do not check populations which the research does not specifically target. For example: a large record review of a diverse population may incidentally include a prisoner or an international citizen, but you should not check those categories if the focus of the study has nothing to do with that status.

Check All That Apply (at least one item must be selected)

### ADDITIONAL INFORMATION:

□ Children (individuals under age 18)

□ Wards of the State (Children)

□ Emancipated Minors

☐ Students

□ College of Medicine Students

□ UK Medical Center Residents or House Officers

□ Impaired Consent Capacity Adults

□ Pregnant Women/Neonates/Fetal Material

□ Prisoners

☐ Non-English Speaking (translated long or short form)

□ International Citizens

□ Normal Volunteers

□ Military Personnel and/or DoD Civilian Employees

Patients

Please visit the <u>IRB Survival Handbook</u> for more information on:

- Children/Emancipated Minors
- Students as Subjects
- Prisoners
- Impaired Consent Capacity Adults
- Economically or Educationally Disadvantaged Persons

Other Resources:

- UKMC Residents or House Officers [see requirement of GME]
- Non-English Speaking [see also the E-IRB Research Description section on this same topic]
- <u>International Citizens</u> [<u>DoD SOP</u> may apply]
- Military Personnel and/or DoD Civilian Employees

### Assessment of the potential recruitment of subjects with impaired consent capacity (or likelihood):

Check this box if your study does NOT involve direct intervention or direct interaction with subjects (e.g., record-review research, secondary data analysis). If there is no direct intervention/interaction you will not need to answer the impaired consent capacity questions.

Does this study focus on adult subjects with any conditions that present a high *likelihood* of impaired consent capacity or *fluctuations* in consent capacity? (see examples below)

Yes ← No

If Yes and you are not filing for exemption certification, go to "Form T", complete the form, and attach it using the button below.

### Examples of such conditions include:

- Traumatic brain injury or acquired brain injury
- Severe depressive disorders or Bipolar disorders
- Schizophrenia or other mental disorders that
- involve serious cognitive disturbances
- Stroke
- Developmental disabilities
- Degenerative dementias
- CNS cancers and other cancers with possible CNS involvement
- Late stage Parkinson's Disease

- Late stage persistent substance dependence
- Ischemic heart disease
- HIV/AIDS
- COPD
- Renal insufficiency
- Diabetes
- Autoimmune or inflammatory disorders
- Chronic non-malignant pain disorders
- Drug effects
- Other acute medical crises

Attachments

### INFORMED CONSENT/ASSENT PROCESS/WAIVER

0 unresolved comment(s)

For creating your informed consent attachment(s), please download the most up-to-date version listed in "All Templates" under the APPLICATION LINKS menu on the left, and edit to match your research project.

### Additional Resources:

- Informed Consent/Assent Website
- Waiver of Consent vs. Waiver of Signatures
- Sample Repository/Registry/Bank Consent Template

### Consent/Assent Tips:

- If you have multiple consent documents, be sure to upload each individually (not all in a combined file).
- If another site is serving as the IRB for the project, attach the form as a "Reliance Consent Form" so the document will not receive a UK IRB approval stamp; the reviewing IRB will need to stamp the consent forms.
- Changes to consent documents (e.g., informed consent form, assent form, cover letter, etc...) should be reflected in a 'tracked changes' version and uploaded separately with the Document Type "Highlighted Changes".
- It is very important that only the documents you wish to have approved by the IRB are attached; DELETE OUTDATED FILES previously approved versions will still be available in Protocol History.
- Attachments that are assigned a Document Type to which an IRB approval stamp applies will be considered the version(s) to be
  used for enrolling subjects once IRB approval has been issued.
   Document Types that do NOT get an IRB approval stamp are:
  - · "Highlighted Changes",
  - · "Phone Script", and
  - "Reliance Consent Form",
  - "Sponsor's Sample Consent Form".

### How to Get the Section Check Mark

- 1. You must:
  - a) provide a response in the text box below describing how investigators will obtain consent/assent, and
  - b) check the box for at least one of the consent items and/or check mark one of the waivers
- 2. If applicable attach each corresponding document(s) as a read-only PDF.
- 3. If you no longer need a consent document approved (e.g., closed to enrollment), or, the consent document submitted does not need a stamp for enrolling subjects (e.g., umbrella study, or sub-study), only select "Stamped Consent Doc(s) Not Needed".
- 4. After making your selection(s) be sure to scroll to the bottom of this section and SAVE your work!



### Check All That Apply-

- □ Informed Consent Form (and/or Parental Permission Form and/or translated short form)
- □ Assent Form
- ☐ Cover Letter (for survey/questionnaire research)
- Phone Script
- Informed Consent/HIPAA Combined Form
- □ Debriefing and/or Permission to Use Data Form
- □ Reliance Consent Form
- □ Sponsor's sample consent form for Dept. of Health and Human Services (DHHS)-approved protocol
- ☐ Stamped Consent Doc(s) Not Needed

### Attachments

| Attach Type | File Name |
|---|---|
| Informed Consent/HIPAA Combined Form | Informed Consent Clean 818.pdf |
| Informed Consent/HIPAA Combined Form | 72601_Stamped Consent Form_551584.pdf |
| Informed Consent/HIPAA Combined Form clean consent 53023.pdf | |
| Phone Script | Phone Consent clean.pdf |

#### **Informed Consent Process:**

Using active voice, describe how investigators will obtain consent/assent. Include:

- the circumstances under which consent will be sought and obtained
- the timing of the consent process (including any waiting period between providing information and obtaining consent)
- · who will seek consent
- · how you will minimize the possibility of coercion or undue influence
- the method used for documenting consent
- if applicable, who is authorized to provide permission or consent on behalf of the subject
- if applicable, specific instruments or techniques to assess and confirm potential subjects' understanding of the information

Note: all individuals authorized to obtain informed consent should be designated as such in the E-IRB "Study Personnel" section of this application.

Special considerations may include:

- · Obtaining consent/assent for special populations such as children, prisoners, or people with impaired decisional capacity
- Research Involving Emancipated Individuals
   If you plan to enroll some or all prospective subjects as emancipated, consult with UK legal counsel prior to submitting this application to the IRB. Include research legal counsel's recommendations in the "Additional Information" section as a separate document
- Research Involving Non-English Speaking Subjects
   For information on inclusion of non-English speaking subjects, or subjects from a foreign culture, see IRB Application Instructions for Recruiting Non-English Speaking Participants or Participants from a Foreign Culture.
- Research Repositories
   If the purpose of this submission is to establish a research repository describe the informed consent process. For guidance regarding consent issues, process approaches, and sample language see the <a href="Sample Repository/Registry/Bank Consent Template">Sample Repository/Registry/Bank Consent Template</a>.

Patient Navigation Arm: Clinic staff will work to identify current diabetic patients who are not compliant with the diabetic standard of care, defined as not having had an appointment with their primary care provider (PCP) within the last 3 months. Clinic staff will contact these patients to inform them of the UK- Faith Moves Mountains Diabetes Research Project. If a patients indicates interest in the program, the clinic staff will inform our research staff. All patients who are interested will be invited to attend a scheduled health screening event. Project staff will administer the informed consent document. Study personnel for all phases of the project will provide a clear explanation of the project and invite questions. Our informed consent forms are written in a basic language. Interested participants will be asked to provide their signature on the informed consent forms. A copy of the signed consent will be provided for all participants. All forms will be read to participants to allay concerns about limited literacy. No non-English speaking or cognitively impaired participants will be recruited.

For the additional interrview with a subset of CCN participants (n=30), We will contact previous CCN participants who have given us permission to recontact them about participation in future related studies. During these conversations, we will use the attached phone script for consent to explain all aspects of participation in the interview and invite the participant to enroll in the study. Throughout this process, participants will be encouraged to ask questions and reminded of their right to discontinue participation at any time. After completing the consent process, participants will be invited to schedule a 60-minute interview.

Clinic Site will work with FMM Project Staff to verify appointments made and/or kept by participants at the conclusion of the 6- week intervention and again at the 3-month milestone. Clinic Site will identify a point of contact/representative for FMM Staff to reach out to in order to verify this information.

If needed, Clinic Site will identify a point of contact/representative for FMM Staff to reach out for scheduling facility usage for the intervention and follow-up sessions.

Participants will be asked to contact the investigator, Dr. Nancy Schoenberg at 859-323-8175 should they have any complaints. If they have any questions about their rights as a volunteer in this research, they will be asked to contact the staff in the Office of Research Integrity at the University of Kentucky at 859-257-9428 or toll free at 1-866-400-9428.

□ Request for Waiver of Informed Consent Process

If you are requesting IRB approval to waive the requirement for the informed consent process, or to alter some or all of the elements of informed consent, complete, Section 1 and Section 2 below.

Note: The IRB does not approve waiver or alteration of the consent process for greater than minimal risk research, except for planned emergency/acute care research as provided under FDA regulations. Contact ORI for regulations that apply to single emergency use waiver or acute care research waiver (859-257-9428).

### **SECTION 1.**

Check the appropriate item:

■I am requesting a waiver of the requirement for the informed consent process.

■I am requesting an alteration of the informed consent process.

If you checked the box for this item, describe which elements of consent will be altered and/or omitted, and ju alteration.

### **SECTION 2.**

Explain how each condition applies to your research.

- a) The research involves no more than minimal risk to the subject.
- b) The rights and welfare of subjects will not be adversely affected.
- c) The research could not practicably be carried out without the requested waiver or alteration.
- d) Whenever possible, the subjects or legally authorized representatives will be provided with additional pertinent information after they have participated in the study.

If you are requesting IRB approval to waive the requirement for signatures on informed consent forms, your research activities must fit into one of three regulatory options:

- 1. The only record linking the participant and the research would be the consent document, and the principal risk would be potential harm resulting from a breach of confidentiality (e.g., a study that involves participants who use illegal drugs).
- 2. The research presents no more than minimal risk to the participant and involves no procedures for which written consent is normally required outside of the research context (e.g., a cover letter on a survey, or a phone script).
- 3. The participant (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm, the research presents no more than minimal risk to the subject, and there is an appropriate alternative mechanism for documenting that informed consent was obtained.

Select the option below that best fits your study.

If the IRB approves a waiver of signatures, participants must still be provided oral or written information about the study. To ensure you include required elements in your consent document, use the **Cover Letter Template** as a guide. There is an <u>English</u> and a <u>Spanish</u> version.



### Option 1

### Describe how your study meets these criteria:

- a) The only record linking the participant and the research would be the consent document:
- b) The principal risk would be potential harm resulting from a breach of confidentiality (i.e., a study that involves subjects who use illegal drugs).

Under this option, each participant (or legally authorized representative) must be asked whether (s)he wants to sign a consent document; if the participant agrees to sign a consent document, only an IRB approved version should be used.

### Option 2

### Describe how your study meets these criteria:

- a) The research presents no more than minimal risk to the participant:
- b) Involves no procedures for which written consent is normally required outside of the research context (i.e. a cover letter on a survey, or a phone script):

### Option 3

### Describe how your study meets these criteria:

- a) The subject (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm.
- b) The research presents no more than minimal risk to the subject.
- c) There is an appropriate alternative mechanism for documenting that informed consent was obtained.

to existing knowledge in this area. For interventional research, search PubMed and ClinicalTriplicgor for duplicative origing and completed high with same condition and intervention(s).
outcomes from TZOM lived we ensuring optimal dirtical care and self-management. Because the previdence of diabetes has tripled since 2005, the already low supply of primary care physicial a the potential or migrating the adventer effects of these a detailed in the case of these a detailed in the case of the case

- Closed Proposed from the whether adjusts of the exponential and whether adjusts of the exponential and whether adjusts of the exponential and whether adjusts of the exponential and the e

ruit subjects. Hease consider the following items and provide additional information as needed so that the IRB can follow each step of the recruitment pro-

- Now will the study team livestry potential pathogoset?
   Will you sub-individuous livestry potential pathogoset?
   Will you sub-individuous livestry and studied in hose?
   Will you sub-individuous livestry li

mation on recruiting and advertising:

RB Application Instructions - Advertisements
 H Guide to Identification and Recruitment of Human Sub

ucky, primally in Leither and Hales Couries. Community perfered reculainest cliens advantages (over direct reculsivers) such as 'entitling hard to reach individuals with impeded access to divice, varieting selection has of healthir periodical belief with a fail and proteinling high direct received by the access and to use of which are the community organizations to determine their interest in periodical and individual belief.

Above Mondayin-MF Framer Francis (and Each of Ex water) to did not not seen a second of third by profing approved bear of specimity digitality Sometring Evers. The Project Dath will consider controlled the limit of the Second Controlled to the International Application of the Second Controlled Co

real Province Perceiones Recombined Service Special RL University of Kentucky Center for Clarical and Transformal Sciences to develop a short video that may be used on social made or showed with potential recombined short. Link: This shumb-based interpretable, Link: This shumb-based interpretable, Link: This shumb-based interpretable, and in the control of the con

# Describe how the research will be condu Perentiate between procedures that involve standardiroutine dinical care and those that will be performed specifically for this Officerate between procedure that in other standard ordinate defined care and took that will be professed upderfloadly be the research project. List medications that are explicitly interesting only a section of permitted during such participants. The received days are designed to receive the received of the received Complete Engineering American a parter agrees to published in the research daily, PAD impost and will inform how shad the dipole by convering and deformers a time to administer informed consent and then classified beautiful based on tomers to desire and the properties of the Complete Brain Science. and Blanch Science. and Blanch Science. and Blanch Science. The Complete Brain Science and the science and the sci ants who chose to participate in the social support survey will complete the one time survey and be comp Attachments Attach Type Data Continues in Persianni Ministeria in Persianni Mi beside the an adulty of the recorded and deplayed of the Targers on government of the Confidence of th Disorbe any priested prise — including physical popular point legal, whiley to reducefly subjects, or other risks. Assess the sentaureses and full code of each mini. Which risks many which a subject is willingues to participate in the study? Disorbeit field, where risks of study, before, otherwise procedures pre-procedure may encounter when the study. Calculation research—causache disclaim and could arise white conducting research in the fall and studyes you may use to handle those shadow. Disorbeit only risks in rights from this. Beards Describe printed first to levels to shotly perinquists—including diagnostic or therepaids, physically applicabilistics, physically perindically considered bearders to shotly perinquistics or the printed by th Describe demands treatments or apportunities that might be available to those who choose not to participate in the study, and which offer the subject equal or greater advantages. If applicable, his should include a depart tecords. Privary, and Confessiolary. Jacoby where the state and the openioness will be stated and how the researcher will ensure the privary and confessiolary of bells. Generally who will have access to the dishabetee Secretary where the immagned share the shody to complete. If data/specimens will be maintained, specify whether identifiers will be removed from the maintained information/material. It identifiers will not be removed, provide justification for relating them and describe how you will prototo confidentially. If the data/specimens will be destroyed, worth that this will not wisher accession and time and will achieve to applicable facility requirements. If applicable, describe procedures for sharing data/specimens with collaborators not affiliated with UK. For additional considerations: Return of Research Results or Incidental Research Findings MH Genomic Data Suss. Dotal Data Two sources of data will be collected; blom-Table 1: Variables Data sources and collector Main outcomes HbA1C, Hood pressure, waist circumference, I Additional outcomes: Sall has a Non outcomes Although Company and well consideration. Bill Project staff Association in regular and proposed staff Association in regular and proposed staff Association in regular and proposed staff and proposed staff Association in regular and proposed staff and proposed staff Association in regular and proposed staff and proposed staff Association in regular and proposed staff and proposed staff Association in regular and proposed staff Association in regular and proposed staff Association in regular and proposed staff Association in regular and proposed staff Confedentially in the proposed staff and association in regular and proposed staff Confedentially being promise prove or unput copy of this with the particular community being variety and proposed staff and association in regular and association in regular and association in r and only all activities of the property of the W. RB colores state that IRB-related research records must be retained for a minimum of 5 years after study closurs. Do you confirm that you will retain all IRB-related rec Periopents will be offered \$35 for each assessment (survey). There will be three assessments over the course of their participation, participants will receive their payment for each assessment. Perioparts in the social support sub-indy will be consented expanding and compensated \$35 for the one time survey. Patient Navigation Arm: FMM will compensate the clinical site in an amount to be negotiated with each site for their participation in the project. A maximum amount will be d Populs a file of services and/or tests that will not be paid for by the sponsor and/or the study (e.g., MPI, HPV, Keep in mind that a subject will not loow what is "standard"—and that for If you are conducting greater than minimal risk research, or your clinical investigation is NE-hunded, describe your Data and Safety Monitoring Plan (DSMP). Click have 5 If this is a non-poressored investigation initiated protocol consistened greater than minimal risk research, and if you are planning on using a Data and Safety Monitoring Data. If the material collected for this study will be used by members of the research team or shared with other researchers for future studies, please address the following: In an interminant consecution for this study was set used by therefore an other research terms of any belief by describe the types, categories and/or purposes of the study research described any time of the additional own described principlyconfederality protection for that will be put into dates described principlyconfederality protection that will be put into dates described principlyconfederality protection of that will be put into dates described principles of time specimensification will be used described procedures for safety precedensification will secondary researchers described the processors, and distribution, whicheased of representations. Fig. the sal-logical generates active information in the sale per condepand specimens will be large. Fig. the sale-logical generates active information in the sale purpose of the face research deviational contents or security as a content of the sale process of the face research deviational contents or security as a content of the sale process of the face research deviational contents or contents or contents of the face research transport or contents of the sale process of the sal Are you recruiting or expect to enroll Non-English Speaking Subjects or Subjects from a Foreign Culture? (does not include short form use for incidentally encountered non-English subjects) This is to be a fine or the subject of th Non-English Speaking Subjects or Subjects from a Foreign Culture Describe how information about the study will be communicated to potential subjects appropriate for their culture, and if necessary, how new information about the research may be relayed to subjects during the study. When recruiting Non-English epeaking subjects, provide a consent documents in the "informed Consent" section. Cultural and Language Consultants: The PI is required to identify someone who is willing to serve as the cultural consultant to the IRB. This person should be findler who to is sitting to serve as the collust gonellast to the IES. This person should be findler with the culture of the subject population and/or be able to verify that translated documents are the equiv This person should be findler with the siding of these any streeted in talk dispraced. See the calculations of the subject population and the street of the IES approach. See the calculations are subject to the subject population of the IES approach. See the calculations are subject to the IES approach to the calculations are subject to the IES approach to the IES approach to the IES approach to the IES approach to the IES approach to IES approach t

Section 10 Page 2 of 4

Local recognitudens:

If you will conduct research at an international location, identify and desce

relevant local regulations

data privacy regulations

applicate laws

children review requirements for human subject protection

Local Requirements:

For more details, see the IRB Application Instructions on Research Involving Non-Ground St.

Flease provide links or sources where possible. If the project has been or will be reviewed by a local ethics review board, attach a copy in the "Additional Infor-

Multilevel linear mixed effects models are used for the continuous outcomes. Models incorporate fixed effects corresponding to trial arm, categorical time, and their interaction, with primary interests described in the next paragraph. To further account for the study design, models incorporate random site effects, random household effects within sites, and an unstructured covariance matrix for repeated measures over time from the same subject. Standard error estimates and degrees of freedom are calculated using the approach of Kenward and Roger (1997).

Analyses are based on intention-to-treat, and utilize all available data. Tests are two-sided at the 5% significance level. Analyses are conducted in SAS Version 9.4 (SAS Institute, Cary, NC).